CLINICAL TRIAL: NCT03645174
Title: Fiberoptic-guided Endotracheal Intubation Through Laryngeal Mask Airway in Manikin; Long Endotracheal Tube vs. Aintree Intubating Catheter
Brief Title: Long Endotracheal Tube vs. Aintree Intubating Catheter for Fiberoptic-guided Intubation in Manikin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, In-kyong Yi, Clinical assitant professor, Ajou University School of Medicine
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AJIRB-MED-OBS-18-226
Record Dates: First submitted 2018-08-22; First posted 2018-08-24 (Actual); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Intubation;Difficult
Keywords: intubation; Aintree; Laryngeal mask airway; fiberoptic

STUDY DESIGN:
Intervention Model Description: Manikin model Intubators are residents of Anesthesiology
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aintree catheter (Active Comparator): Fiberoptic-guided intubation through LMA, using Aintree catheter
  Interventions: Device: Aintree catheter
- Long tube (Experimental): Fiberoptic-guided intubation through LMA, using long tube
  Interventions: Device: Using long tube

INTERVENTIONS:
Device: Using long tube — Fiberoptic-guided intubation through LMA, using long tube
  Arms: Long tube
Device: Aintree catheter — Fiberoptic-guided intubation through LMA, using Aintree catheter
  Arms: Aintree catheter

SUMMARY:
In difficult airway situation, fiberoptic-guided endotracheal intubation through laryngeal mask airway(LMA) is one of option. Aintree catheter is a device to help change LMA to endotracheal tube, but it needs complex and multiple process. Long endotracheal tube can solve this problem of Aintree catheter. The purpose of this study is proving the efficacy of long endotracheal tube compared to Aintree cathter in fiberoptic-guided intubation through LMA.

DETAILED DESCRIPTION:
In difficult aiway situation, fiberoptic-guided endotracheal intubation through laryngeal mask airway(LMA) is one of option according to Difficult intubation guidelines. First, insert LMA and insert fiberoptic through LMA. Second, insert endotracheal tube using fiberoptic as a guide. This process has several problem. Removal of LMA is impossible, so there is a risk of dislodging of endotracheal tube.

Aintree catheter is developed to this problem. Insert Aintree catheter through LMA using fiberoptic, and remove LMA, finally insert endotracheal tube throug Aintree catheter. But the problem of this method is that the whole process is complex and takes long time. And there is a risk of impeding of endotracheal tube at glottis level because the difference of diameters between endotracheal tube and aintree catheter.

Long endotracheal tube could solve the problems mentioned above. Through LMA, insert endotracheal tube using fiberoptic as a guide. Tube is long enough to remove LMA without a risk of dislodging. And after removal of LMA, tube can be cut for optimizing length.

So the purpose of this study is comparing the efficacy of Aintree catheter method and Long tube method in manikin.

ELIGIBILITY:
Inclusion Criteria:

* Residents of Anesthesiology
* Who has less than 10 times of experience of fiberoptic intubation

Exclusion Criteria:

* Who has more than 10 times of experience of fiberoptic intubation
* Who deny participating in the study

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-01-15 (Actual)

PRIMARY OUTCOMES:
Intubation time | 3 minutes
  from entry of fiberoptic at LMA to Ambu bagging

SECONDARY OUTCOMES:
Success rate | 5 minutes
  Failure is esophageal intubation or disloding of endotracheal tube in any process
Difficulty score | 5 minutes
  Subjective score using numeric rating scale (1; extremely easy - 10; extremely difficult)

CONTACTS AND LOCATIONS:
Overall Officials: In Kyong Yi, MD, Principal Investigator — Ajou University School of Medicine
Locations (1):
- Ajou university school of medicine, Suwon, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No
only for personally requested

REFERENCES:
- [Derived] Chae YJ, Lee H, Jun B, Yi IK. Conversion of I-gel to definitive airway in a cervical immobilized manikin: Aintree intubation catheter vs long endotracheal tube. BMC Anesthesiol. 2020 Jun 18;20(1):152. doi: 10.1186/s12871-020-01069-9. PMID 32552828